CLINICAL TRIAL: NCT04565184
Title: Monitoring the Effectiveness and Safety of Artesunate-Amodiaquine and Artemether-Lumefantrine During the Treatment of Uncomplicated Plasmodium Falciparum Malaria Among Children in Yaounde, Cameroon
Brief Title: Effectiveness and Safety of Artesunate-Amodiaquine and Artemether-Lumefantrine for the Treatment of Malaria in Yaounde
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Yaounde 1 (Other)
Collaborators: Malaria Research Capacity Development in West and Central Africa Consortium (Unknown); Developing Excellence in Leadership, Training and Science Africa Initiative (Unknown); Wellcome Trust (Other); United Kingdom Department for International Development (Unknown)
Responsible Party: Principal Investigator, Professor Wilfred Fon Mbacham, Principal Investigator, University of Yaounde 1
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MARCAD/UYI/NPTN/12/16
Record Dates: First submitted 2020-09-17; First posted 2020-09-25 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Malaria,Falciparum
Keywords: Malaria; Plasmodium falciparum; Artesunate-amodiaquine; Artemether-lumefantrine; Effectiveness; Safety
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: Eligible children for whom parent/guardian informed consent are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) in the ratio 1:1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Artesunate-amodiaquine (Arm A) (Experimental): Artesunate-amodiaquine (Coarsucam®: Sanofi-Aventis, France) is co-packaged as artesunate 50 mg and amodiaquine hydrochloride USP equivalent to amodiaquine base of 153.1 mg. Each child shall be given one, two or three tablets depending on the weight.
  Interventions: Drug: Artesunate-amodiaquine combination
- Artemether-lumefantrine (Arm B) (Active Comparator): Artemether-lumefantrine (Coartem®: Novartis, Switzerland) is formulated as tablets and will be provided in blister packs. Each tablet contains 20 mg artemether and 120 mg lumefantrine. Every pack has a picture showing how the drug should be given and contains two blisters for each day with one, two or three tablets depending on the weight of the child.
  Interventions: Drug: Artemether, Lumefantrine Drug Combination

INTERVENTIONS:
Drug: Artesunate-amodiaquine combination — Artesunate-amodiaquine (Coarsucam®: Sanofi-Aventis, France) is co-packaged as artesunate 50 mg and amodiaquine hydrochloride USP equivalent to amodiaquine base of 153.1 mg. Each child shall be given one, two or three tablets depending on the weight.
  Other Names: Coarsucam
  Arms: Artesunate-amodiaquine (Arm A)
Drug: Artemether, Lumefantrine Drug Combination — Artemether-lumefantrine (Coartem®: Novartis, Switzerland) is formulated as tablets and will be provided in blister packs. Each tablet contains 20 mg artemether and 120 mg lumefantrine. Every pack has a picture showing how the drug should be given and contains two blisters for each day with one, two or three tablets depending on the weight of the child
  Other Names: Coartem®
  Arms: Artemether-lumefantrine (Arm B)

SUMMARY:
Artesunate-amodiaquine and artemether-lumfantrine are currently being used for the treatment of uncomplicated Plasmodium falciparum in Cameroon. Globally, many studies have reported high efficacy and safety of artemisinin-based combination therapies (ACTs) mostly under strict supervision of drug intake and limited to children less than 5 years of age. Patients over 5 years of age are usually not involved in such studies. The main objective of this study is to assess the genetic markers of antimalarial drug resistance and drug metabolism subsequent to the efficacy and safety of artesunate-amodiaquine and artemether-lumefantrine during a 28-day follow-up period in children with acute uncomplicated P. falciparum malaria in Yaounde, Cameroon. A randomized, open-labelled, controlled clinical trial comparing artesunate-amodiaquine (ASAQ) and artemether-lumefantrine (AL) will be carried out from 9th May 2019 to 30th November 2020 at two secondary health centres (Cité Verte and Minkoameyos) in Yaounde. The study participants shall include febrile patients aged 6 months to 10 years, with confirmed uncomplicated P. falciparum infection. Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) in the ratio 1:1. A minimum sample of 76 patients will be required for the study. With a 20 % increase to allow loss to follow-up and withdrawals during the 28-day follow-up period, 92 patients will be enrolled for each of the two study arms. The study will recruit a total of 184 patients. Drug intake will be partially supervised only for the first dose and subsequent doses administered unsupervised as pertains in routine practice in the field. Patients or their parents/guardians will be advised on the time and mode of administration for the 3 days (D0, D1 and D2) treatment unobserved at home. Follow-up visits will be performed on days 3, 7, 14, 21, and 28 to evaluate clinical and parasitological resolution of their malaria episode as well as adverse events. Polymerase chain reaction (PCR) genotyping of merozoite surface proteins 1 and 2 (msp-1, msp-2) as well as glutamate rich protein (GLURP) will be used to differentiate between recrudescence and new infection.

DETAILED DESCRIPTION:
Background: Artesunate-amodiaquine and artemether-lumfantrine are currently being used for the treatment of uncomplicated Plasmodium falciparum in Cameroon. Globally, many studies have reported high efficacy and safety of artemisinin-based combination therapies (ACTs) mostly under strict supervision of drug intake and limited to children less than 5 years of age. Patients over 5 years of age are usually not involved in such studies.

Objective: To assess the genetic markers of antimalarial drug resistance and drug metabolism subsequent to the efficacy and safety of artesunate-amodiaquine and artemether-lumefantrine during a 28-day follow-up period in children with acute uncomplicated P. falciparum malaria in Yaounde, Cameroon.

Study sites: District Hospital Cité Verte and District Medical Centre Minkoa Meyos in Yaounde, Cameroon. The two drugs, artesunate-amodiaquine and artemether-lumefantrine will be tested in each site.

Study period: 9th May 2019 to 30th November 2020.

Study design: This surveillance study is a two-arm, open-label, randomized controlled clinical trial.

Patient population: Febrile patients aged 6 months to 10 years, with confirmed uncomplicated P. falciparum infection. Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) in the ratio 1:1.

Sample size: A minimum sample of 76 patients will be required for the study. With a 20 % increase to allow loss to follow-up and withdrawals during the 28-day follow-up period, 92 patients will be enrolled for each of the two study arms. The study will recruit a total of 184 patients.

Treatment (s) and follow-up: Drug intake will be partially supervised only for the first dose and subsequent doses administered unsupervised as pertains in routine practice in the field. Patients or their parents/guardians will be advised on the time and mode of administration for the 3 days (D0, D1 and D2) treatment unobserved at home. Follow-up visits will be performed on days 3, 7, 14, 21, and 28 to evaluate clinical and parasitological resolution of their malaria episode as well as adverse events. Polymerase chain reaction (PCR) genotyping of merozoite surface proteins 1 and 2 (msp-1, msp-2) as well as glutamate rich protein (GLURP) will be used to differentiate between recrudescence and new infection.

Classification of treatment outcomes Classification of treatment outcomes will be done based on the WHO 2009 guidelines: treatment failure (Early Treatment Failure-ETF, Late Clinical failure-LCF and Late Parasitological Failure-LPF) and treatment success (Adequate Clinical and Parasitological Response-ACPR).

ELIGIBILITY:
Inclusion Criteria:

* Children of either gender, aged 6 months to 120 months will be recruited.
* Acute uncomplicated P. falciparum malaria confirmed by microscopy using Giemsa-stained thick film with an asexual parasite density within the range 1000 to 200000 parasites/μl.
* Presenting with fever (axillary temperature ≥ 37.5oC) or having a history of fever in the preceding 24 hours.
* Able to ingest tablets orally (either suspended in water or uncrushed with food).
* Willing to participate in the study with written informed consent from parent/guardian.
* Willing and able to attend the clinic on stipulated regular follow-up visits.

Exclusion Criteria:

* Mixed with another Plasmodium species detected by microscopy.
* Children who are currently suffering or had the following within the last 2 months: tuberculosis, HIV, schistosomiasis, diabetes mellitus, cardiovascular disease, gout, rheumatoid arthritis, underlying chronic hepatic or renal disease, hypoglycaemia, jaundice, respiratory distress, and other inflammatory related diseases.
* Signs/symptoms indicating severe/complicated malaria" according to WHO criteria (WHO definition) such as:

Not able to drink or breast feed. Persistent vomiting (>2 episodes within previous 24 hours). Convulsions (>1 episode within previous 24 hours). Lethargic/unconscious. Severe anaemia (haemoglobin < 5 g/dl).

* Serious gastrointestinal disease.
* Presence of severe malnutrition defined as a child aged between 6-60 months whose weight-for-high is below -3 z-score (W/H < 70%) or has symmetrical edema involving at least the feet or has a mid-upper arm circumference < 115 mm).
* Regular medication, which may interfere with anti-malarial pharmacokinetics.
* History of hypersensitivity reactions or contraindications to any of the medicine (s) being tested or used as alternative treatment (s).
* Individuals who have taken part in anti-malarial efficacy and safety studies in the last 3 months.
* Participants who have taken anti-malarial drugs in the last one month.

Ages: 6 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 242 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment success and adverse events following treatment with artesunate-modiaquine and artemether-lumefantrine during 28 days follow-up period in children with acute uncomplicated P. falciparum malaria in Yaounde | 18 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) and follow-up will be done for a duration of 28 days.

SECONDARY OUTCOMES:
Proportion of patients with early treatment failure, late clinical failure, late parasitological failure or an adequate clinical and parasitological response as indicators of efficacy according to the WHO 2009 guidelines | 18 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) and follow-up will be done for a duration of 28 days. Recrudescence will be distinguished from re-infection by polymerase chain reaction (PCR) analysis
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 18 months
  Eligible children for whom parent/guardian informed consents are obtained will be randomized to receive either artesunate-amodiaquine (group A) or artemether-lumefantrine (group B) and follow-up will be done for a duration of 28 days.
Number of children with single nucleotide polymorphisms of P. falciparum genes responsible for AS-AQ and AL resistance | 18 months
  Pre-treatment and recrudescence/reinfection samples during follow-up shall be used to characterize the molecular markers of Plasmodium falciparum chloroquine resistant transporter(Pfcrt), Plasmodium falciparum multi-drug resistant 1 (Pfmdr1), and Plasmodium falciparum K13 (Pfk13) propellar domain conferring resistance to artemisinins or partner drugs.
Number of children haboring single nucleotide polymorphisms in key genes involved in the metabolism of AS-AQ and AL | 18 months
  Pre-treatment samples shall be used to characterize the human pharmacogenomic biomarkers (N-acetyl transferase 2-NAT2 and cytochrome P450: CYP2A6, CYP2B6, CYP2C8, CYP2C9, CYP2C19, CYP3A4, and CYP3A5)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred Fon Mbacham, PhD, Principal Investigator — Biotechnology Centre, University of Yaounde I
Locations (1):
- District Medical Center Minkoa Meyos, Yaoundé, Center, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
Research findings will be communicated with the scientific community and policymakers. This will be done through public engagements and publications in peer-review journals.
Supporting Information: Study Protocol, CSR
Time Frame: 30th November 2020 for at least 10 years
Access Criteria: Not available for now

REFERENCES:
- [Derived] Niba PTN, Nji AM, Ali IM, Akam LF, Dongmo CH, Chedjou JPK, Fomboh CT, Nana WD, Oben OLA, Selly-Ngaloumo AA, Moyeh MN, Ngu JA, Ludovic AJ, Aboh PM, Ambani MCE, Omgba PAM, Kotcholi GB, Adzemye LM, Nna DRA, Douanla A, Ango Z, Ewane MS, Ticha JT, Tatah FM, Dinza G, Ndikum VN, Fosah DA, Bigoga JD, Alifrangis M, Mbacham WF. Effectiveness and safety of artesunate-amodiaquine versus artemether-lumefantrine for home-based treatment of uncomplicated Plasmodium falciparum malaria among children 6-120 months in Yaounde, Cameroon: a randomized trial. BMC Infect Dis. 2022 Feb 21;22(1):166. doi: 10.1186/s12879-022-07101-2. PMID 35189818